CLINICAL TRIAL: NCT05791981
Title: Multi-site Feasibility and Acceptability of a Faith-based Mind-body Intervention for Black Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-1023; NCI-2023-02353 (Other: NCI-CTRP Clinical Trials Registry); R01AT012375 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Psychosocial; Mind-body

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harmony & Health Intervention (Group 1) (Experimental): Participants randomized to the Harmony and Health intervention group will attend group-based in-person intervention sessions at FOP or COGIC. on.
  Interventions: Behavioral: Harmony & Health Intervention; Device: Fitbit
- Attention Control (Group 2) (Experimental): Participants randomized to the attention control condition will participate in in-person group-based health education sessions twice a week for 8 weeks with a trained interventionist and will receive 4 monthly newsletters (20 total contacts).
  Interventions: Behavioral: Attention Control; Device: Fitbit

INTERVENTIONS:
Behavioral: Harmony & Health Intervention — Participants will attend group in person sessions 2 times each week for 8 weeks. The sessions will be 45 minutes long. In each session, there will be an introduction, 30 minutes of gentle yoga-based poses and breathing exercises, and then 10 minutes of guided relaxation and scripture meditation.
  Participants will be instructed to practice the exercises at home 2 times each week during the entire 6-month period. You will be given instructions and a yoga mat, belt, and block. After your Week 9 assessment, you will attend in-person or Zoom sessions 1 time each month over the final 4 months of the study
  Arms: Harmony & Health Intervention (Group 1)
Behavioral: Attention Control — Participants will attend group in-person health education sessions 2 times each week for 8 weeks. The sessions will be 45 minutes long and will include discussions of disease prevention and other health and well-being topics. After your Week 9 assessment, you will have the ability to attend additional in-person or Zoom health education sessions 1 time each month over the final 4 months of the study.
  Arms: Attention Control (Group 2)
Device: Fitbit — Participants will be given a Fitbit and instructions on how to use it. The Fitbit will record your physical activity and report it to the study staff.

SUMMARY:
To test a program that combines yoga and Christian spirituality (called Harmony & Health) to learn if it can help participants exercise more.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of this multi-site, community-based, two-arm randomized controlled feasibility trial is to evaluate the feasibility of recruitment, retention, and adherence to the HH intervention and attention control conditions and acceptability of assessments across sites. Black adults who are insufficiently active will be randomized to the HH intervention or an attention control group. We hypothesize that we will meet our recruitment goal of 50 participants per site (10 participants per month), >80% of participants will be retained at post-intervention and follow-up, and >80% will adhere to sessions. After follow-up, we will conduct interviews with community partners (n=2), delivery agents (n=2), and participants (n=20) at each site (N=44 total) to assess acceptance and refine training and implementation protocols in preparation for a future large-scale multi-site randomized controlled trial to test the efficacy of HH.

Secondary Objectives:

Secondary objectives include assessing changes in sitting time, physical activity, and psychosocial wellbeing from baseline to post-intervention as defined below.

1. Sitting time. Sitting time will be measured using an activPAL, a small and slim thigh-worn device that directly measures postural aspects of sedentary behavior (e.g., sitting, lying down, upright), and provides time spent sitting and bouts. Additionally, self-reported sedentary behavior will be assessed via the Sedentary Behavior Questionnaire.
2. Physical activity. Physical activity will be measured using an activPAL, a small and slim thigh-worn device that directly measures steps and intensity-specific physical activity duration. Additionally, self-reported physical activity will be assessed via the Godin Leisure-Time Exercise Questionnaire.
3. Psychosocial wellbeing. Psychosocial wellbeing, including perceived stress, depressive symptoms, and quality of life, will be assessed using the 10-item Perceived Stress Scale (PSS), Center for Epidemiologic Studies Depression Scale (CES-D), and SF-36 Short Form Health Survey.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age
2. Self-identify as Black or African American
3. Able to read, speak, and write in English
4. Self-report doing <90 minutes/week of physical activity
5. Self-report sitting ≥6 hours/day
6. Body mass index [BMI] ≥25.0 kg/m2 based on self-reported height and weight
7. Able to provide informed consent
8. Able to pass the Physical Activity Readiness Questionnaire (PARQ) or provide physician's clearance to participate

Exclusion Criteria:

1. <18 years of age
2. Does not identify as Black or African American
3. Unable or uncomfortable participating in English
4. Self-reports doing ≥90 minutes/week of physical activity
5. Self-reports sitting for <6 hours/day
6. BMI <25.0 kg/m2
7. Absolute contraindications to unassisted physical activity based on the PARQ (e.g., acute MI, orthopedic and musculoskeletal limitations)
8. Practicing yoga or enrolled in another program targeting physical activity, sitting time, or weight loss
9. Pregnant or planning to become pregnant during the 6 month study period
10. Planning to move from the Houston or Northeast Texas areas during the 6 month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity of training and implementation across sites | 6 months
  Fidelity will be achieved if there is ≥90% adherence to intervention delivery and receipt.

CONTACTS AND LOCATIONS:
Overall Officials: Scherezade Mama, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org